CLINICAL TRIAL: NCT03875859
Title: A Phase 2 Open Label, Single Arm Trial to Investigate the Efficacy and Safety of Topical Remetinostat Gel as Neoadjuvant Therapy in Patients Undergoing Surgical Resection of Squamous Cell Carcinoma (SCC)
Brief Title: Topical Remetinostat Gel as Neoadjuvant Therapy in Patients With Squamous Cell Carcinoma (SCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The available study medication reached expiry (logistics).
Sponsor: Kavita Sarin (Other)
Collaborators: Medivir (Industry)
Responsible Party: Sponsor-Investigator, Kavita Sarin, Assistant Professor of Dermatology., Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-49542; SKIN0050 (Other: OnCore)
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — remetinostat

STUDY DESIGN:
Intervention Model Description: Open label, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Remetinostat (Experimental): Subjects will apply remetinostat gel 1% to at least 1 SCC: Topical remetinostat gel 1% applied 3 times daily.
  Interventions: Drug: Remetinostat

INTERVENTIONS:
Drug: Remetinostat — Topical 1% remetinostat gel
  Other Names: suberohydroxamic acid phenyl ester (SHAPE); SHAPE Gel;; SHP-141;; and 4-[[8-(hydroxyamino)-1,8-dioxooctyl]oxy]-benzoic acid methyl ester

SUMMARY:
The primary purpose of this study is to determine if 8 weeks of topical remetinostat applied three times daily will suppress Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
The primary purpose of this study is:

* to determine if 8 weeks of topical remetinostat gel applied 3 times daily (TID) under occlusion will suppress SCC growth
* to determine the overall response rate (ORR) of SCCs after 8 weeks of treatment with topical remetinostat gel 1%, as measured by at least 30% decrease in greatest area (in mm2).

  * Subjects with at least 1 biopsy-proven cutaneous SCC will be recruited for this study.
  * Subjects will apply remetinostat gel 1% to at least 1 SCC.
  * Non-invasive cutaneous SCC lesions, including Bowen's disease, are also eligible for this study
  * There is 1 treatment option: Topical remetinostat gel 1% applied 3 times daily.
  * The study is a single arm, open label design
  * For purposes of ClinicalTrials.gov, there is no secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Must have at least one biopsy-proven cutaneous SCC or SCC in situ (SCC-IS) lesion greater than or equal to 5 mm. Non-invasive SCC lesion(s), including Bowen's disease (SCC-IS), are eligible, but must be amenable to surgical resection.
2. 18 years of age or older.
3. Must be willing to apply the topical remetinostat 3 times daily for 8 weeks and cover with an occlusive bandage.
4. Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months)
5. Sexually active women of child bearing potential (WCBP) and male patients with a female partner of child-bearing potential must agree to use acceptable methods of contraception to avoid pregnancy (for example, oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) before the first dose of study therapy and for 3 months after the last dose of study therapy
6. Has signed and dated the current, approved informed consent document.

Exclusion Criteria:

1. Any large (> 20 mm) SCC lesion. Patients with large SCC lesion(s) will be referred for evaluation for surgical resection.
2. Inoperable locally-advanced and/or non-cutaneous metastatic SCC.
3. SCC lesion(s) in cosmetically-sensitive areas (e.g. tip of nose, eyelid) are not eligible for enrollment. (If a patient has SCC lesion(s) in other areas, those tumor(s) may be considered for enrollment.)
4. Taking any medication known to affect SCC growth
5. Within the past 6 months, has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study. Specifically, these include the topical use at the site of the study tumors:

   * Glucocorticoids
   * Retinoids either systemically or topically at the tumor site (e.g., etretinate, isotretinoin, tazarotene, tretinoin, adapalene)
   * Alpha-hydroxy acids (e.g., glycolic acid, lactic acid) to the tumor site
   * 5-fluorouracil or imiquimod
6. Has received treatment with systemic chemotherapy within 60 days prior to starting study medication.
7. Currently receiving systemic medications that could affect SCC tumors (e.g., oral retinoids) or might interact with remetinostat
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, recurrent seizure history or psychiatric illness/social situations that would limit compliance with study requirements.
9. Moderate to significant immunosuppression (e.g., active cancer, significant autoimmune disease) and/or receiving immunosuppressive drugs that result in moderate to significant immunosuppression (e.g. low dose oral glucocorticoids do not necessarily exclude a patient)
10. Known or previous hypersensitivity to HDACi
11. History of congestive heart failure, cardiac arrhythmias, or other findings of ventricular dysfunction.
12. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Y Sarin, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remetinostat
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Remetinostat
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR)
Description: Overall response (OR) will be assessed in squamous cell carcinoma (SCC). Objective response (OR) will defined as the number of lesions with either a complete response (CR) or a partial response (PR) among all eligible and treated lesions, any time within 10 weeks.
  * Complete Response (CR) = Disappearance of target lesion
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesion
  * Overall Response (OR) = CR + PR
Time Frame: 10 weeks
Population: All treated lesions for all participants were included in the analysis.
Measure: Number; unit: tumor lesions
Arm/Group | Remetinostat
Number analyzed (Participants) | 4
tumor lesions
  CR | 5
  PR | 0
  OR | 5

2. Secondary Outcome: Adverse Events Contributing to Treatment Discontinuation or Interruption
Description: Adverse events (AEs) contributing to treatment discontinuation or interruption are reported as the number of such events, a number without dispersion.
Time Frame: 8 weeks
Measure: Number; unit: adverse events
Arm/Group | Remetinostat
Number analyzed (Participants) | 4
adverse events | 1

3. Secondary Outcome: Participants Who Discontinued Treatment or Had Treatment Interruption
Description: The number of participants who discontinued treatment or experienced treatment interruption within the first 8 weeks of treatment are reported as the number of such participants, a number without dispersion.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Remetinostat
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Remetinostat
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remetinostat (N=4)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT03875859/Prot_SAP_000.pdf